CLINICAL TRIAL: NCT05680480
Title: A Phase Ⅱ, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Telitacicept in Lupus Nephritis
Brief Title: A Study of Telitacicept in Lupus Nephritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18C030
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Lupus Nephritis
Keywords: lupus; nephritis; Telitacicept; RC 18
MeSH Terms: conditions — Lupus Nephritis; Nephritis | interventions — telitacicept; RC-18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telitacicept 240 mg (Experimental): Telitacicept 240 mg given SC weekly plus standard therapy through week 48.
  Interventions: Biological: Telitacicept 240 mg
- Telitacicept 160 mg (Experimental): Telitacicept 160 mg given SC weekly plus standard therapy through week 48.
  Interventions: Biological: Telitacicept 160 mg
- Placebo (Placebo Comparator): Placebo given SC weekly plus standard therapy through week 48.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Telitacicept 240 mg — Participants will receive Telitacicept 240mg weekly in addition to SOC for 48 weeks.
  Other Names: RC18 240 mg
  Arms: Telitacicept 240 mg
Biological: Telitacicept 160 mg — Participants will receive Telitacicept 160mg weekly in addition to SOC for 48 weeks.
  Other Names: RC18 160 mg
  Arms: Telitacicept 160 mg
Drug: Placebo — Participants will receive placebo weekly in addition to SOC for 48 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Telitacicept in adult patients with active lupus nephritis.

DETAILED DESCRIPTION:
This is a phase 2, multicentre, randomised, double-blind, placebo-controlled study to evaluate the efficacy and safety of telitacicept versus placebo while taking standard of care (SOC) treatment in adult subjects with active proliferative lupus nephritis (LN).

ELIGIBILITY:
Main Inclusion Criteria:

1. Males or females aged 18-75 years of age, inclusive.
2. Diagnosis of systemic lupus erythematosus according to American College of Rheumatology criteria (1997).
3. Active, biopsy-proven proliferative lupus nephritis Class III or IV with/without the presence of Class V, or pure Class V according to the 2003 ISN/RPS classification. The renal biopsy must be performed within 1 year prior to the screening visit or during screening period. The biopsy report will be used to confirm subject eligibility.
4. Positive serum antibody results, defined as positive anti-nuclear antibody (ANA) and/or a positive anti-dsDNA serum antibody based on the study's central laboratory results.
5. Active renal disease at screening requiring induction therapy with high dose corticosteroids (HDCS) with mycophenolate mofetil (MMF) or other oral forms of mycophenolate.
6. Induction therapy for active renal disease: HDCS with mycophenolate mofetil (MMF) or other oral forms of mycophenolate should be initiated within 60 days prior to or on Day 1 (baseline). Initiation of induction is when both HDCS and MMF have been started.
7. Able to understand the requirements of the study and provide written informed consent.

Main Exclusion Criteria:

1. Known hypersensitivity or contraindication to any drug products they plan to receive (e.g., MMF, corticosteroids).
2. History of allergy to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
3. Received any of the following therapies:

   1. Treatment with any B cell targeted therapy (e.g., rituximab), unless it can be shown that B cells have returned to baseline level or normal;
   2. Received tumor necrosis factor inhibitors, interleukin receptor blockers, or other small molecules or biologics (including Belimumab) during the 12 weeks prior to screening or the 5 half-lives of the drug, whichever is longer;
   3. Received any experimental drugs during the 12 weeks prior to screening or the 5 half-lives of the drug, whichever is longer;
   4. Received plasma separation or plasma exchange during the 6 weeks prior to screening;
   5. Subjects who required dialysis within 1 year prior to screening.
   6. Received a live vaccine or live-attenuated vaccine within 4 weeks prior to screening or expected to vaccinate during the study.
   7. Received BCG Vaccine within 1 year prior to screening.
4. History of severe active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident, cerebritis, or CNS vasculitis) requiring intervention within 60 days of baseline (Day 1).
5. History of a major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant or are due to receive transplantation.
6. Significant, unstable or uncontrolled acute or chronic diseases not due to SLE (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy, or infectious diseases) which, in the opinion of the principal investigator, could confound the results of the study or put the subject at undue risk.
7. Plan to undergo surgery or have any medical disease, laboratory abnormality, or condition that, in the opinion of the principal investigator, makes the subject unsuitable for the study.
8. History of drug or alcohol abuse or dependence within 364 days prior to baseline (Day 1).
9. Nursing or pregnant female, or male or female who prepared for parenthood during the study.
10. History of malignant tumors within the last 5 years, excluding adequately treated skin cancer (basal or squamous cell) or carcinoma in situ of cervix.
11. Have acute or chronic infection requiring treatment.
12. HIV positive.
13. Hepatitis B: Patients positive for HBsAg are excluded; Patients negative for HBsAg but positive for Anti-HBc, regardless of Anti-HBs antibody status, will require test for HBV DNA: if HBV DNA positive, patients will be excluded; if HBV DNA negative, patients will be eligible to enroll.
14. Hepatitis C antibody positive.
15. History of COVID-19 within 4 weeks prior to screening or history of hospitalization due to severe Covid-19 within 12 months prior to screening.
16. eGFR<30 mL/min/1.73 m2 using CKD-EPI.
17. Renal biopsy showed 50% glomerulosclerosis.
18. Have a Grade 3 or greater laboratory abnormality based on the Adverse Event Severity Grading Tables.
19. Subjects who in the opinion of the investigator are not suitable to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Complete Renal Response (CRR) | Week 48
  CRR is defined as estimated glomerular filtration rate (GFR) is no more than 20% below the baseline value or ≥ 60 mL/min/1.73m^2 and 24-hour urinary protein: creatinine ratio ≤ 0.5 mg/mg and did not receive prohibited or rescue therapy resulting in treatment failure.

SECONDARY OUTCOMES:
Percentage of participants with Partial Renal Response (PRR) | Week 24 and Week 48
  PRR is defined as 24-hour urinary protein: creatinine ratio reduced by 50% compared to baseline value.
Incidence of AE, SAE | Up to Week 48
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A SAE is any untoward medical occurrence that at any dose resulting in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant and which the investigator regards as serious based on appropriate medical judgment.

CONTACTS AND LOCATIONS:
Locations (45):
- China (45):
  - The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Hospital Affiliated to the Army Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Liuzhou Workers' Hospital, Liuchow, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Handan First Hospital, Handan, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The Third Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Northern Theater Command of the Chinese People's Liberation Army, Shenyang, Liaoning
  - The Affiliated Hospital of Qinghai University, Xining, Qinghai
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - People's Hospital of Sichuan Province, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Fourth Affiliated Hospital, Zhejiang University School of Medicine, Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397